CLINICAL TRIAL: NCT01004302
Title: Ventral Capsular/Ventral Striatal Gamma Capsulotomy for Obsessive-compulsive Disorder: a Randomized Controlled Trial
Brief Title: Radiosurgical Treatment for Obsessive-compulsive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Our Co sources were in a state of advanced decay. That prolonged our surgical procedures, making them inconveniently and perhaps dangerously long (> 12 hours)
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAPPesq 521/02; CAPPesq 0968/05; CONEP 4891
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Obsessive-compulsive Disorder
Keywords: Obsessive-compulsive disorder; Radiosurgery; Psychosurgery; Treatment outcome; Randomized Controlled Trials
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Radiosurgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham surgery (Sham Comparator)
  Interventions: Procedure: ventral capsular/ventral striatal gamma capsulotomy
- Active radiosurgery (Active Comparator)
  Interventions: Procedure: ventral capsular/ventral striatal gamma capsulotomy

INTERVENTIONS:
Procedure: ventral capsular/ventral striatal gamma capsulotomy — Comparison of active radiosurgical with sham radiosurgeries
  Other Names: Gamma ventral capsulotomy; Anterior capsulotomy; Gamma Knife radiosurgery

SUMMARY:
Up to 40% of Obsessive-Compulsive Disorder (OCD) patients do not respond to conventional treatments (medications or behavior therapy). For some of them, a neurosurgical treatment can be indicated. Among various surgical techniques, Gamma Knife radiosurgery has the advantage of not requiring the production of burr hole openings in the skull. However, there are no randomized controlled trials of radiosurgical procedures.

The investigators' aim is to investigate whether radiosurgery for the treatment of severe and refractory OCD is efficacious and safe, by a double-blind, randomized controlled trial. Forty-eight refractory OCD patients will be randomized into two different groups: the first one will receive standard radiosurgery; the second group will be submitted to a false radiosurgery ("sham operation"). Patients who had been previously submitted to sham surgery will be able to undergo real operations after one year of follow-up, when blinding is broken. For a minimum period of one year, patients will be periodically followed-up in terms of psychiatric changes (including OCD symptoms), global functioning, cognitive/personality changes and neuroimaging findings.

DETAILED DESCRIPTION:
Various studies have demonstrated that good treatment responses in Obsessive Compulsive Disorder (OCD) are often obtained in 60 to 80 % of patients, whether employing serotonin reuptake inhibitors or behavior therapy. However, a subgroup of OCD patients are refractory to the classical therapeutic options, even after maximum dosage regimens and sufficiently long treatment follow-ups are devised. Severe psychosocial and occupational impairments are meanwhile observable. These subjects are often referred to stereotactic neurosurgeries. Among the various surgical techniques, a radiosurgical modality (double-shot ventral capsular/ventral striatal - VC/VS gamma capsulotomy, or simply double-shot gamma ventral capsulotomy) has been recently developed. On the other hand, there are no randomized controlled trials of Gamma Knife radiosurgeries in Psychiatry.

The aim of this study is to investigate whether double-shot VC/VS gamma capsulotomy is efficacious and to describe its adverse events/complications profiles, in a double-blind, randomized controlled trial of this radiosurgical technique for the treatment of refractory OCD.

Forty-eight refractory OCD patients will be randomized into two different groups: the first one will receive standard radiosurgery; the second group will be submitted to a false radiosurgical intervention ("sham operation"). All subjects will be previously assessed by a preliminary clinical/psychiatric interview, as well as by extensive specific instruments regarding psychiatric diagnosis, OCD evolution and severity, anxiety/depression symptoms, tics expression, psychosocial impairment, personality changes, etc. A neuropsychological tests battery will also be employed. All patients will be offered a periodical follow-up, during which assessment scales and neuroimaging exams (magnetic resonance imaging) will be repeated. Patients who had been previously submitted to placebo surgery will be able to undergo real operations after the one-year follow-up period, when blinding is broken. Scores results will be analyzed among the groups, as well as adverse events profiles, cognitive/personality changes, clinical global functioning and neuroimaging findings. Improvements in Yale-Brown Obsessive Compulsive Scale (YBOCS) and Clinical Global Impression (CGI) scores will be taken as the primary treatment response criteria.

ELIGIBILITY:
Inclusion Criteria:

* A DSM-IV diagnosis of OCD as the main diagnostic entity. If comorbid axis I or II disorders are present, OCD symptoms are the most troublesome among disorders.
* Age range between 18 and 60 years old.
* At least 5 years of OCD symptoms.
* "Yale-Brown Obsessive-Compulsive Scale" (YBOCS) scores greater than 26 (or greater than 13, for isolated obsessions or compulsions).
* Refractoriness criteria fulfilled.
* To be accepted by the "best estimate" method as a treatment refractory patient. It consists in the careful examination of each patient's history by two OCD specialists, so as to confirm refractoriness status.

Refractoriness criteria:

* At least 3 serotonin reuptake inhibitors have been tried before (selective or not). One of these trials must have included clomipramine. All drugs were used for a minimum of 12 weeks, at the maximum doses or the maximally tolerated doses.
* Previous participation in a cognitive behavior therapy program (exposure and response prevention), for a minimum of 20 hours' time; or participation for some time, without subsequent adherence, due to severe OCD symptoms, and acceptance of the independent review board.
* YBOCS scores reductions after adequate drug therapy and psychotherapy not better than 25 %, or confirmation of no clinical improvements by the mental health professionals who were responsible for the treatments of the patient.
* By the end of adequately conducted pharmacological trials, "Clinical Global Impression" (CGI) scores not better than minimal improvement.
* Previous use of at least two antidepressant augmentation strategies (such as the association of a typical or atypical antipsychotic, another serotonin reuptake inhibitor, a benzodiazepine, lithium carbonate, or buspirone), in adequate doses for a sufficient period of time, without satisfactory responses.

Exclusion Criteria:

* Less than 18 years or more than 60 years of age.
* Past history of head injury, with posttraumatic amnesia.
* Past or general medical condition, or neurological illness with brain compromise (severe and in active phase)
* History of physiological effects of a substance, as determinant of psychopathological symptoms, or cumulative signs of alcohol or drug abuse in the Central Nervous System (such cortical atrophy), confirmed by a neuroimaging scan.
* Pregnancy or lactation.
* Refusal to participate in radiosurgical procedures.
* Refusal to sign the Patient Information and Consent Form, or refusal to take part in this study.
* History of mental retardation and/or being unable to understand the Patient Information and Consent Form, confirmed by poor performance on neuropsychological tests.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2003-07; Primary Completion 2013-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
A reduction of at least 35 % in the Yale-Brown Obsessive Compulsive Scale (YBOCS) scores and an "improved" or "much improved" score on the Clinical Global Impression (CGI) scale | One year

CONTACTS AND LOCATIONS:
Overall Officials: Antonio C Lopes, MD, PhD, Principal Investigator — Department and Institute of Psychiatry, General Hospital, University of São Paulo Medical School
Locations (1):
- Department and Institute of Psychiatry, General Hospital, University of São Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Batistuzzo MC, Hoexter MQ, Taub A, Gentil AF, Cesar RC, Joaquim MA, D'Alcante CC, McLaughlin NC, Canteras MM, Shavitt RG, Savage CR, Greenberg BD, Noren G, Miguel EC, Lopes AC. Visuospatial Memory Improvement after Gamma Ventral Capsulotomy in Treatment Refractory Obsessive-Compulsive Disorder Patients. Neuropsychopharmacology. 2015 Jul;40(8):1837-45. doi: 10.1038/npp.2015.33. Epub 2015 Feb 3. PMID 25645373
- [Derived] Lopes AC, Greenberg BD, Canteras MM, Batistuzzo MC, Hoexter MQ, Gentil AF, Pereira CA, Joaquim MA, de Mathis ME, D'Alcante CC, Taub A, de Castro DG, Tokeshi L, Sampaio LA, Leite CC, Shavitt RG, Diniz JB, Busatto G, Noren G, Rasmussen SA, Miguel EC. Gamma ventral capsulotomy for obsessive-compulsive disorder: a randomized clinical trial. JAMA Psychiatry. 2014 Sep;71(9):1066-76. doi: 10.1001/jamapsychiatry.2014.1193. PMID 25054836